CLINICAL TRIAL: NCT04932200
Title: A Prospective Multicenter Cohort Study on the Timing of Emergency Endoscopy for Esophagogastric Variceal Bleeding in Cirrhosis
Brief Title: The Timing of Emergency Endoscopy for Esophagogastric Variceal Bleeding in Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Collaborators: Beijing Friendship Hospital (Other); The First Affiliated Hospital of Nanchang University (Other); Fudan University (Other); Southwest Hospital, China (Other); Beijing Shijitan Hospital, Capital Medical University (Other); Fuyang NO.2 Renmin Hospital (Unknown); Hubei Hospital of Traditional Chinese Medicine (Other); Wuhan No.1 Hospital (Other); Wuhan Puren Hospital (Other); Tianyou Hospital Affiliated to Wuhan University of Science and Technology (Other); The Central Hospital of Enshi Tujia And Miao Autonomous Prefecture (Other); Yichang Central People's Hospital (Other); Shiyan Renmin Hospital (Unknown); Hanyang University (Other); The Third People's Hospital of Hubei Province (Other); Chibi Renmin Hospital (Unknown)
Responsible Party: Principal Investigator, ChenMingkai, Professor, Renmin Hospital of Wuhan University
Other Study IDs: WDRY2021-K061
Record Dates: First submitted 2021-06-11; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Liver Cirrhosis; Portal Hypertension; Esophageal Varix Bleeding
Keywords: esophagogastric variceal bleeding; emergency endoscopy; timing
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- urgent-endoscopy group: the time interval from gastroenterologic consultation to the start of emergency endoscopy < 6 hours
- early-endoscopy group: the time interval from gastroenterologic consultation to the start of emergency endoscopy between 6 and 24 hours

SUMMARY:
This study is a prospective, multi-center and observational clinical study. Investigators would like to explore the optimal emergency endoscopy timing in cirrhosis patients with esophagogastric variceal bleeding (EGVB) by evaluating and comparing the efficacy and safety of emergency endoscopy performed at different times ( within 6 hours or between 6 and 24 hours after gastroenterologic consultation ) and its impact on the short-term prognosis.

DETAILED DESCRIPTION:
Between July 2021 and April 2022, patients with cirrhosis undergoing emergency endoscopy due to EGVB are enrolled consecutively according to the following criteria: (1) age≥18 years; (2) A definite diagnosis of cirrhosis (confirmed by medical history, laboratory examination and imaging examination); (3) The cause of bleeding was identified as esophageal and/or gastric vein rupture. Exclusion criteria are as follows: (1) End-stage diseases of major organs (such as heart failure, chronic obstructive pulmonary disease, end-stage renal disease, and malignancies other than hepatocellular carcinoma); (2) The subject (or legal representative/guardian) refused to sign the informed consent.

Patients were divided into urgent-endoscopy group (< 6h) and early-endoscopy group (6h-24h) according to the time interval from gastroenterologic consultation to the start of emergency endoscopy.

Investigators will collect patients' data of baseline character, treatment, postoperative and follow-up. All patients will be followed up until death or the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years
* A definite diagnosis of cirrhosis (confirmed by medical history, laboratory examination and imaging examination)
* The cause of bleeding was identified as esophageal and/or gastric vein rupture

Exclusion Criteria:

* End-stage diseases of major organs (such as heart failure, chronic obstructive pulmonary disease, end-stage renal disease, and malignancies other than hepatocellular carcinoma)
* The subject (or legal representative/guardian) refused to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cirrhosis undergoing emergency endoscopy due to EGVB are enrolled this study.
Sampling Method: Non-Probability Sample
Enrollment: 608 (Estimated)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
six-week mortality rate | 6 weeks after treatment
  Patients died in six weeks after emergency endoscopy due to rebleeding or other complications associated with cirrhosis.

SECONDARY OUTCOMES:
Immediate success hemostasis rate | within 24 hours after traetment
  Successful immediate hemostasis refers to successful hemostasis under endoscopy, and no active bleeding manifestations such as hematemesis, hemorrhagic shock and progressive decline of hemoglobin within 24 hours.
five-day rebleeding rate | 5 days after treatment
  Patients rebleeded due to esophageal and gastric varices bleeding in five days after treatment.
detection rate of bleeding site | during endoscopy
  Identify the site of bleeding during endoscopy.
mean operating time | during endoscopy
  The time interval between the beginning and end of endoscopy.
the needs of salvage treatment | 6 weeks
  Salvage treatment refers to the additional three-chamber and two-capsule compression hemostasis, re-endoscopic therapy, interventional therapy or surgical treatment due to failure of hemostasis by emergency endoscopy or re-bleeding after successful hemostasis.

CONTACTS AND LOCATIONS:
Overall Officials: Mingkai Chen, PHD, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garcia-Tsao G, Abraldes JG, Berzigotti A, Bosch J. Portal hypertensive bleeding in cirrhosis: Risk stratification, diagnosis, and management: 2016 practice guidance by the American Association for the study of liver diseases. Hepatology. 2017 Jan;65(1):310-335. doi: 10.1002/hep.28906. Epub 2016 Dec 1. No abstract available. PMID 27786365
- [Background] Tripathi D, Stanley AJ, Hayes PC, Patch D, Millson C, Mehrzad H, Austin A, Ferguson JW, Olliff SP, Hudson M, Christie JM; Clinical Services and Standards Committee of the British Society of Gastroenterology. U.K. guidelines on the management of variceal haemorrhage in cirrhotic patients. Gut. 2015 Nov;64(11):1680-704. doi: 10.1136/gutjnl-2015-309262. Epub 2015 Apr 17. PMID 25887380
- [Background] Reiberger T, Puspok A, Schoder M, Baumann-Durchschein F, Bucsics T, Datz C, Dolak W, Ferlitsch A, Finkenstedt A, Graziadei I, Hametner S, Karnel F, Krones E, Maieron A, Mandorfer M, Peck-Radosavljevic M, Rainer F, Schwabl P, Stadlbauer V, Stauber R, Tilg H, Trauner M, Zoller H, Schofl R, Fickert P. Austrian consensus guidelines on the management and treatment of portal hypertension (Billroth III). Wien Klin Wochenschr. 2017 Nov;129(Suppl 3):135-158. doi: 10.1007/s00508-017-1262-3. Epub 2017 Oct 23. PMID 29063233
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines for the management of patients with decompensated cirrhosis. J Hepatol. 2018 Aug;69(2):406-460. doi: 10.1016/j.jhep.2018.03.024. Epub 2018 Apr 10. No abstract available. PMID 29653741
- [Background] Cheung J, Soo I, Bastiampillai R, Zhu Q, Ma M. Urgent vs. non-urgent endoscopy in stable acute variceal bleeding. Am J Gastroenterol. 2009 May;104(5):1125-9. doi: 10.1038/ajg.2009.78. Epub 2009 Mar 31. PMID 19337243
- [Background] Hsu YC, Chung CS, Tseng CH, Lin TL, Liou JM, Wu MS, Hu FC, Wang HP. Delayed endoscopy as a risk factor for in-hospital mortality in cirrhotic patients with acute variceal hemorrhage. J Gastroenterol Hepatol. 2009 Jul;24(7):1294-9. doi: 10.1111/j.1440-1746.2009.05903.x. PMID 19682197
- [Background] Chen PH, Chen WC, Hou MC, Liu TT, Chang CJ, Liao WC, Su CW, Wang HM, Lin HC, Lee FY, Lee SD. Delayed endoscopy increases re-bleeding and mortality in patients with hematemesis and active esophageal variceal bleeding: a cohort study. J Hepatol. 2012 Dec;57(6):1207-13. doi: 10.1016/j.jhep.2012.07.038. Epub 2012 Aug 8. PMID 22885718
- [Background] Jung DH, Huh CW, Kim NJ, Kim BW. Optimal endoscopy timing in patients with acute variceal bleeding: A systematic review and meta-analysis. Sci Rep. 2020 Mar 4;10(1):4046. doi: 10.1038/s41598-020-60866-x. PMID 32132589
- [Background] Lau JYW, Yu Y, Tang RSY, Chan HCH, Yip HC, Chan SM, Luk SWY, Wong SH, Lau LHS, Lui RN, Chan TT, Mak JWY, Chan FKL, Sung JJY. Timing of Endoscopy for Acute Upper Gastrointestinal Bleeding. N Engl J Med. 2020 Apr 2;382(14):1299-1308. doi: 10.1056/NEJMoa1912484. PMID 32242355
- [Background] Huh CW, Kim JS, Jung DH, Yang JD, Nam SW, Kwon JH, Kim BW. Optimal endoscopy timing according to the severity of underlying liver disease in patients with acute variceal bleeding. Dig Liver Dis. 2019 Jul;51(7):993-998. doi: 10.1016/j.dld.2019.01.013. Epub 2019 Jan 29. PMID 30803858